CLINICAL TRIAL: NCT05706402
Title: A Double-Blind Randomized Controlled Trial of N-acetylcysteine (NAC) for the Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: N-acetylcysteine (NAC) for the Treatment of Acute Exacerbation of COPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok Wang Chun, Clinical Assistant Professor, Honorary Specialist, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 22-710
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: N-acetylcysteine; Chronic Obstructive Pulmonary Disease; Chronic Obstructive Pulmonary Disease exacerbation; Clinical trial
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This study is a double-blind randomised controlled trial on NAC as an adjunctive treatment for acute COPD exacerbation. The randomization will be done via computer software with half of the patients randomized to received oral NAC (600 mg twice daily) and half receive placebo, with randomization ratio being 1 to 1. Patients in the two randomised group will be asked to participate in the study for a maximum of 1 week.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcysteine (Experimental)
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Patients will be randomized to receive oral N-acetylcysteine at 600 mg twice daily for 1 week. The randomization will be done via computer software with half of the patients randomized to receive NAC. Patients will also be given standard treatment for your COPD exacerbation and can continue the use of usual inhalers for COPD.
  Arms: N-acetylcysteine
Drug: Placebo — Patients will be randomized to receive placebo for 1 week. The randomization will be done via computer software with half receive placebo. Patients will also be given standard treatment for your COPD exacerbation and can continue the use of usual inhalers for COPD.
  Arms: Placebo

SUMMARY:
Patients with Chronic obstructive pulmonary disease (COPD) experience gradually deteriorating lung function, which may be complicated by acute exacerbations. N- acetylcysteine (NAC) is frequently used in patients with COPD as a mucolytic. Besides its mucolytic effects, high-dose NAC has additional benefits in patients with stable COPD, including improving lung function and reducing exacerbations. Studies on the dose-dependent effects of NAC in COPD patients showed a high dose of NAC was needed to achieve its antioxidant effects and clinical benefits in COPD patients, whereas a dose of 600 mg once daily was not able to increase glutathione levels. According to a study conducted in Hong Kong on patients with stable COPD, 1 year of treatment with high-dose NAC at 600 mg twice daily improved small airways function in terms of forced expiratory flow and forced oscillation technique, and also significantly reduced exacerbation frequency with a decreasing trend in admission rate. In a meta-analysis, patients treated with NAC had significantly and consistently fewer exacerbations of COPD. The role of NAC was examined in a Delphi consensus study involving 53 COPD experts from 12 countries. Respondents agreed that regular treatment with mucolytic agents could effectively decrease the frequency of exacerbations and the duration of mild-to-moderate exacerbations, while delaying the time to first exacerbation and increasing symptom-free time in COPD patients. The panel also approved the doses of NAC with favourable side effect profiles to be recommended for regular use in patients with a bronchitic phenotype.

However, there have been conflicting results regarding the efficacy of NAC for treating acute exacerbation of COPD. NAC has not been included as an adjunct for the treatment of COPD exacerbation in international guidelines. As NAC is relatively low cost, readily available, and has a favourable side effect profile as a treatment for COPD exacerbation, it is important to properly assess the clinical benefits of NAC as an adjunct to standard medical treatments to hasten recovery. This study is a double-blind randomised controlled trial on NAC as an adjunctive treatment for acute COPD exacerbation. It will assess the role of NAC in the treatment of acute COPD exacerbation.

DETAILED DESCRIPTION:
The aim of the study is to assess the role of NAC in the treatment of acute COPD exacerbation in terms of clinical, physiological, and laboratory parameters, including PaO2, PaO2/FiO2 ratio, PaCO2, SaO2, end tidal CO2, length of stay, coughing, wheezing, dyspnoea, need for supplemental oxygen sputum volume, FEV1, and blood inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40 years or above, either male or female.
2. Patients who are current or ex-smokers

   * Ever-smoker is defined as having smoked at least one cigarette, pipe, water pipe, cigars, or hand rolled cigarettes a day for 1 or more years.
3. Patients with a pre-existing diagnosis of COPD admitted to the general medical and respiratory subspecialty wards for acute COPD exacerbation

   * COPD is defined as dyspnoea and/or chronic productive cough with spirometry confirmation of persistent airflow limitation at FEV1/FVC less than 70%.
   * COPD acute exacerbation is defined as an acute increase in symptoms (one or more of the following: cough frequency and severity, sputum production, dyspnoea) beyond normal day-to-day variations leading to a change in medication.
4. Patients who consent to join this clinical trial

Exclusion Criteria:

1. Patients who are on long-term NAC treatment
2. Patients who are not able to take NAC including drug allergy
3. Patients with other co-existing respiratory diseases including but not limited to asthma, interstitial lung diseases, and bronchiectasis
4. Patients on non-invasive or invasive mechanical ventilation where oral medication is not allowed
5. Patients on long term macrolide treatment
6. Patients on macrolide as antibiotics for COPD exacerbation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The difference in mean PaO2 and the change of PaO2 | day 7; from day 0 to day 7
  The co-primary endpoint of interest is the difference in mean PaO2 on day 7 of treatment and the change of PaO2 from day 0 to day 7.

SECONDARY OUTCOMES:
The change in PaO2/FiO2 ratio | from baseline to day 7
  The change in PaO2/FiO2 ratio from baseline to day 7
The change in sputum volume | from baseline to day 7
  The change in sputum volume on days 4 and 7
The Change in COPD Assessment Test (CAT) score | from baseline to day 7
  The change in CAT score on days 4 and 7. CAT score has a scoring range of 0 to 40. Higher scores indicating the COPD has a greater impact on overall health outcome.
The Change in Leicester cough questionnaire (LCQ) score | from baseline to day 7
  The change in LCQ score on days 4 and 7. The LCQ is assessing 3 domains (physical, psychological and social). The total score range is 3-21 and domain scores range from 1-7. Higher scores indicates a better quality of life.
The Change in the grade of wheeze assessment (Grading system) | from baseline to day 7
  The change in grade of wheeze on days 4 and 7. Grade of wheeze, to be assessed by the PI or Co-I, is a simple bedside assessment can that can assess the severity of COPD. This could allow a simple assessment of the respiratory status for the patients with COPD exacerbation. There will be 3 grades; higher grade indicates a more severe respiratory symptoms.
The change in grade of dyspnoea on the modified Medical Research Council (mMRC) Dyspnoea Scale | from baseline to day 7
  The change in grade of dyspnoea on the modified Medical Research Council (mMRC) Dyspnoea Scale on days 4 and 7. The mMRC scale ranges from grade 0 to 4. Higher grade indicates a higher degree of baseline functional disability due to dyspnoea.
The change in FEV1 | from baseline to day 7
  The change in FEV1 on days 4 and 7
The change in end tidal CO2 | from baseline to day 7
  The change in end tidal CO2 on days 4 and 7
The change in SaO2 | from baseline to day 7
  The change in SaO2 on days 4 and 7
The change in PaCO2 | from baseline to day 7
  The change in PaCO2 on day 7
The time to wean off supplemental oxygen | from baseline to day 7
The length of stay | from baseline to day 7
The blood inflammatory markers | from baseline to day 7
  Blood inflammatory markers including white cell count, neutrophil count, erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), and high-sensitivity CRP (hs-CRP) will also be measured, total 20 mL of blood will be taken. Blood inflammatory markers including white cell count, neutrophil count, ESR, CRP, and hs-CRP will be measured on days 4 and 7. The blood tests arranged for the patients are the basic blood tests for clinical management of COPD exacerbation and it does not involve extra blood testing for the patients.
The 28- and 90-day mortality | from baseline to 28- and 90-day

CONTACTS AND LOCATIONS:
Overall Officials: Wang Chun Kwok, MBBS, Principal Investigator — Division of Respiratory Medicine, Department of Medicine, The University of Hong Kong, Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwok WC, Chan SKS, Chiang KY, Ho CMJ. A double-blind randomized controlled trial of N-acetylcysteine (NAC) for the treatment of acute exacerbation of chronic obstructive pulmonary disease. Respirol Case Rep. 2024 Aug 6;12(8):e01449. doi: 10.1002/rcr2.1449. eCollection 2024 Aug. PMID 39108325